CLINICAL TRIAL: NCT06095817
Title: Continuity of Military Transition Study: Project VALOR
Brief Title: Project VALOR: Veteran Stress and Wellbeing
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding to continue
Sponsor: Cornell University (Other)
Collaborators: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Smithers2023
Record Dates: First submitted 2023-10-18; First posted 2023-10-23 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Alcohol Use Disorder; Depression
Keywords: Alcohol-Related Disorders; Anxiety; Alcoholism; Self Medication; Stress Disorders, Post-Traumatic; Depression; Psychological Distress; Drinking Behavior; Substance-Related Disorders
MeSH Terms: conditions — Alcoholism; Depression; Alcohol-Related Disorders; Anxiety Disorders; Stress Disorders, Post-Traumatic; Drinking Behavior; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: One group will receive an opportunity to engage with a personalized internet-delivered brief intervention (IDBI) and the second group will not be granted access. This IDBI will serve as a second booster intervention for half o those randomized into the treatment condition. For the other half randomized into the treatment condition, this IDBI will serve as an initial intervention coming 12 months after separation from the military.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Condition (Experimental): Participants assigned to the intervention condition will be invited to engage with an internet-based intervention at the start of the study (12 months following their separation)
  * Half of those in the intervention condition will have already received two prior IDBIs (as part of the DoD funded study) within the first 6 months of separation.
  * The other half of those in the intervention condition will have received no prior IDBIs.
  Interventions: Behavioral: Internet Delivered Brief Intervention (IDBI)
- Control (No Intervention): The control group will not be offered this month-12 internet-based intervention.
  * Half of those in the control condition will have received two earlier IDBIs (as part of the DoD funded study) within the first 6 months of their separation.
  * The other half of those in the control condition will have received no prior IDBIs.

INTERVENTIONS:
Behavioral: Internet Delivered Brief Intervention (IDBI) — The intervention is an online module that can be accessed through smartphone, tablet, computer or other device. Participants will receive information about alcohol expectancies, alcohol use and norms, identity (service member, veteran, civilian), sleep, stress, and strategies for coping on the job.
  Arms: Intervention Condition

SUMMARY:
This study will examine the efficacy of an internet-based brief intervention designed to reduce risky behavior veterans as the move into their second year post-Army. Up to 350 veterans drawn from The Network Study (Dept of Defense; Award number: W81XWH1920001) will be recruited with the intention of drawing a final sample of 300. Study participants will be randomly assigned to either the intervention or the control group, stratified by age and gender.

DETAILED DESCRIPTION:
The combination of alcohol use and negative emotional states is a particularly toxic combination for suicide risk. The current study examines changes in alcohol/drug use/misuse and depression as veterans transition further into their post-Army environment and offers a personalized internet-based brief intervention intended to prevent/reduce alcohol misuse and depression in this population.

The study's objectives are to empirically quantify the form of changes that occur with respect to alcohol use and depression as veterans move into their second year post-Army; to identify stable individual risk factors (e.g., personality, military experiences) and dynamic risk factors (e.g., changes in stressors and normative contexts over time) that may be associated with differential temporal patterns of suicide-related behavior (i.e., alcohol use/misuse) and cognition (i.e., depression); and lastly, to determine whether a simple, internet-delivered brief intervention shown can reduce risky behavior in the veteran population.

ELIGIBILITY:
Inclusion Criteria:

* Is US Army veteran who participated in The Network Study (Dept of Defense; Award number: W81XWH1920001)
* Seeks/engages in civilian employment
* Lives in US

Exclusion Criteria:

* Retired with no plans to seek civilian employment
* Living outside of the US
* Separated from the National Guard or Reserves

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-10-06 (Actual)

PRIMARY OUTCOMES:
Change in Heavy Episodic Drinking | Through study completion, data collected quarterly from 15 to up to 24 months post-separation from the Army
  Single Alcohol Screening Question (SASQ) (Williams and Vinson, 2001)
Change in Modal alcohol consumption | Through study completion, data collected quarterly from 15 to up to 24 months post-separation from the Army
  Daily Drinking Questionnaire (DDQ) (Collins, Parks, & Marlatt, 1985)
Change in Negative Emotional State -- Depression | Through study completion, data collected quarterly from 15 to up to 24 months post-separation from the Army
  The Patient Health Questionnaire (PHQ)-9

SECONDARY OUTCOMES:
Change in Alcohol-related problems | Through study completion, data collected quarterly from 15 to up to 24 months post-separation from the Army
  Short Rutgers Alcohol Problems Index (S-RAPI) (Earleywine, LaBrie & Pedersen)
Change in Suicidal ideation | Through study completion, data collected quarterly from 15 to up to 24 months post-separation from the Army
  Suicide ideation measure developed by Nock, 2007

OTHER OUTCOMES:
Change in Employment | Through study completion, data collected quarterly from 15 to up to 24 months post-separation from the Army
  Current job situation/Change employment

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Bacharach, PhD, Principal Investigator — Cornell University
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Williams R, Vinson DC. Validation of a single screening question for problem drinking. J Fam Pract. 2001 Apr;50(4):307-12. PMID 11300981
- [Background] Collins RL, Parks GA, Marlatt GA. Social determinants of alcohol consumption: the effects of social interaction and model status on the self-administration of alcohol. J Consult Clin Psychol. 1985 Apr;53(2):189-200. doi: 10.1037//0022-006x.53.2.189. No abstract available. PMID 3998247
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Nock MK, Banaji MR. Prediction of suicide ideation and attempts among adolescents using a brief performance-based test. J Consult Clin Psychol. 2007 Oct;75(5):707-15. doi: 10.1037/0022-006X.75.5.707. PMID 17907852
- [Background] Saunders JB, Aasland OG, Babor TF, de la Fuente JR, Grant M. Development of the Alcohol Use Disorders Identification Test (AUDIT): WHO Collaborative Project on Early Detection of Persons with Harmful Alcohol Consumption--II. Addiction. 1993 Jun;88(6):791-804. doi: 10.1111/j.1360-0443.1993.tb02093.x. PMID 8329970
- [Background] Forbes D, Alkemade N, Mitchell D, Elhai JD, McHugh T, Bates G, Novaco RW, Bryant R, Lewis V. Utility of the Dimensions of Anger Reactions-5 (DAR-5) scale as a brief anger measure. Depress Anxiety. 2014 Feb;31(2):166-73. doi: 10.1002/da.22148. Epub 2013 Jun 25. PMID 23801571
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Britt TW, Adler AB, Sawhney G, Bliese PD. Coping Strategies as Moderators of the Association Between Combat Exposure and Posttraumatic Stress Disorder Symptoms. J Trauma Stress. 2017 Oct;30(5):491-501. doi: 10.1002/jts.22221. PMID 29078001
- [Background] Carver CS. You want to measure coping but your protocol's too long: consider the brief COPE. Int J Behav Med. 1997;4(1):92-100. doi: 10.1207/s15327558ijbm0401_6. PMID 16250744
- [Background] Sayer NA, Frazier P, Orazem RJ, Murdoch M, Gravely A, Carlson KF, Hintz S, Noorbaloochi S. Military to civilian questionnaire: a measure of postdeployment community reintegration difficulty among veterans using Department of Veterans Affairs medical care. J Trauma Stress. 2011 Dec;24(6):660-70. doi: 10.1002/jts.20706. Epub 2011 Dec 7. PMID 22162082
- [Background] Lindgren KP, Neighbors C, Teachman BA, Wiers RW, Westgate E, Greenwald AG. I drink therefore I am: validating alcohol-related implicit association tests. Psychol Addict Behav. 2013 Mar;27(1):1-13. doi: 10.1037/a0027640. Epub 2012 Mar 19. PMID 22428863
- [Background] Grant VV, Stewart SH, O'Connor RM, Blackwell E, Conrod PJ. Psychometric evaluation of the five-factor Modified Drinking Motives Questionnaire--Revised in undergraduates. Addict Behav. 2007 Nov;32(11):2611-32. doi: 10.1016/j.addbeh.2007.07.004. Epub 2007 Jul 13. PMID 17716823
- [Background] Ames GM, Grube JW. Alcohol availability and workplace drinking: mixed method analyses. J Stud Alcohol. 1999 May;60(3):383-93. doi: 10.15288/jsa.1999.60.383. PMID 10371267
- [Background] Ames GM, Grube JW, Moore RS. Social control and workplace drinking norms: a comparison of two organizational cultures. J Stud Alcohol. 2000 Mar;61(2):203-19. doi: 10.15288/jsa.2000.61.203. PMID 10757130
- [Background] Baer JS, Stacy A, Larimer M. Biases in the perception of drinking norms among college students. J Stud Alcohol. 1991 Nov;52(6):580-6. doi: 10.15288/jsa.1991.52.580. PMID 1758185
- [Background] Treloar H, Martens MP, McCarthy DM. The Protective Behavioral Strategies Scale-20: improved content validity of the Serious Harm Reduction subscale. Psychol Assess. 2015 Mar;27(1):340-6. doi: 10.1037/pas0000071. Epub 2015 Jan 5. PMID 25558969
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Hughes ME, Waite LJ, Hawkley LC, Cacioppo JT. A Short Scale for Measuring Loneliness in Large Surveys: Results From Two Population-Based Studies. Res Aging. 2004;26(6):655-672. doi: 10.1177/0164027504268574. PMID 18504506
- [Background] Brown DW, Balluz LS, Heath GW, Moriarty DG, Ford ES, Giles WH, Mokdad AH. Associations between recommended levels of physical activity and health-related quality of life. Findings from the 2001 Behavioral Risk Factor Surveillance System (BRFSS) survey. Prev Med. 2003 Nov;37(5):520-8. doi: 10.1016/s0091-7435(03)00179-8. PMID 14572437
- [Background] Bliese PD, Wright KM, Adler AB, Cabrera O, Castro CA, Hoge CW. Validating the primary care posttraumatic stress disorder screen and the posttraumatic stress disorder checklist with soldiers returning from combat. J Consult Clin Psychol. 2008 Apr;76(2):272-81. doi: 10.1037/0022-006X.76.2.272. PMID 18377123
- [Background] Rehm J, Greenfield TK, Walsh G, Xie X, Robson L, Single E. Assessment methods for alcohol consumption, prevalence of high risk drinking and harm: a sensitivity analysis. Int J Epidemiol. 1999 Apr;28(2):219-24. doi: 10.1093/ije/28.2.219. PMID 10342682
- [Background] Nock MK, Holmberg EB, Photos VI, Michel BD. Self-Injurious Thoughts and Behaviors Interview: development, reliability, and validity in an adolescent sample. Psychol Assess. 2007 Sep;19(3):309-17. doi: 10.1037/1040-3590.19.3.309. PMID 17845122
- [Background] Nock MK, Hwang I, Sampson NA, Kessler RC. Mental disorders, comorbidity and suicidal behavior: results from the National Comorbidity Survey Replication. Mol Psychiatry. 2010 Aug;15(8):868-76. doi: 10.1038/mp.2009.29. Epub 2009 Mar 31. PMID 19337207
- [Background] Norman SB, Schmied E, Larson GE. Predictors of continued problem drinking and substance use following military discharge. J Stud Alcohol Drugs. 2014 Jul;75(4):557-66. doi: 10.15288/jsad.2014.75.557. PMID 24988254
- [Background] Conner KR, Bagge CL, Goldston DB, Ilgen MA. Alcohol and suicidal behavior: what is known and what can be done. Am J Prev Med. 2014 Sep;47(3 Suppl 2):S204-8. doi: 10.1016/j.amepre.2014.06.007. PMID 25145740
- [Background] Neighbors C, Lewis MA, Atkins DC, Jensen MM, Walter T, Fossos N, Lee CM, Larimer ME. Efficacy of web-based personalized normative feedback: a two-year randomized controlled trial. J Consult Clin Psychol. 2010 Dec;78(6):898-911. doi: 10.1037/a0020766. PMID 20873892
- [Background] Cosper R. Drinking as conformity; a critique of sociological literature on occupational differences in drinking. J Stud Alcohol. 1979 Sep;40(9):868-91. doi: 10.15288/jsa.1979.40.868. PMID 513778
- [Background] Holahan CJ, Moos RH, Holahan CK, Cronkite RC. Resource loss, resource gain, and depressive symptoms: a 10-year model. J Pers Soc Psychol. 1999 Sep;77(3):620-9. doi: 10.1037//0022-3514.77.3.620. PMID 10510511
- [Background] Brenner LA, Barnes SM. Facilitating treatment engagement during high-risk transition periods: a potential suicide prevention strategy. Am J Public Health. 2012 Mar;102 Suppl 1(Suppl 1):S12-4. doi: 10.2105/AJPH.2011.300581. Epub 2012 Jan 25. No abstract available. PMID 22390585
- [Background] Kapur N, While D, Blatchley N, Bray I, Harrison K. Suicide after leaving the UK armed forces--a cohort study. PLoS Med. 2009 Mar 3;6(3):e26. doi: 10.1371/journal.pmed.1000026. PMID 19260757
- [Background] Karlamangla A, Zhou K, Reuben D, Greendale G, Moore A. Longitudinal trajectories of heavy drinking in adults in the United States of America. Addiction. 2006 Jan;101(1):91-9. doi: 10.1111/j.1360-0443.2005.01299.x. PMID 16393195
- [Background] Sher L, Braquehais MD, Casas M. Posttraumatic stress disorder, depression, and suicide in veterans. Cleve Clin J Med. 2012 Feb;79(2):92-7. doi: 10.3949/ccjm.79a.11069. PMID 22301558
- [Background] Thomas JL, Wilk JE, Riviere LA, McGurk D, Castro CA, Hoge CW. Prevalence of mental health problems and functional impairment among active component and National Guard soldiers 3 and 12 months following combat in Iraq. Arch Gen Psychiatry. 2010 Jun;67(6):614-23. doi: 10.1001/archgenpsychiatry.2010.54. PMID 20530011
- [Background] Finley EP, Bollinger M, Noel PH, Amuan ME, Copeland LA, Pugh JA, Dassori A, Palmer R, Bryan C, Pugh MJ. A national cohort study of the association between the polytrauma clinical triad and suicide-related behavior among US Veterans who served in Iraq and Afghanistan. Am J Public Health. 2015 Feb;105(2):380-7. doi: 10.2105/AJPH.2014.301957. PMID 25033126
- [Background] Cooper ML, Russell M, Skinner JB, Frone MR, Mudar P. Stress and alcohol use: moderating effects of gender, coping, and alcohol expectancies. J Abnorm Psychol. 1992 Feb;101(1):139-52. doi: 10.1037//0021-843x.101.1.139. PMID 1537960
- [Background] Carver CS, Scheier MF. Situational coping and coping dispositions in a stressful transaction. J Pers Soc Psychol. 1994 Jan;66(1):184-95. doi: 10.1037//0022-3514.66.1.184. PMID 8126648
- [Background] MacLean MG, Lecci L. A comparison of models of drinking motives in a university sample. Psychol Addict Behav. 2000 Mar;14(1):83-7. doi: 10.1037//0893-164x.14.1.83. PMID 10822750
- [Background] CONGER JJ. Alcoholism: theory, problem and challenge. II. Reinforcement theory and the dynamics of alcoholism. Q J Stud Alcohol. 1956 Jun;17(2):296-305. No abstract available. PMID 13336262
- [Background] Frone MR. Are work stressors related to employee substance use? The importance of temporal context assessments of alcohol and illicit drug use. J Appl Psychol. 2008 Jan;93(1):199-206. doi: 10.1037/0021-9010.93.1.199. PMID 18211145
- [Background] Hassija CM, Jakupcak M, Maguen S, Shipherd JC. The influence of combat and interpersonal trauma on PTSD, depression, and alcohol misuse in U.S. Gulf War and OEF/OIF women veterans. J Trauma Stress. 2012 Apr;25(2):216-9. doi: 10.1002/jts.21686. PMID 22522738
- [Background] Jones E, Fear NT. Alcohol use and misuse within the military: a review. Int Rev Psychiatry. 2011 Apr;23(2):166-72. doi: 10.3109/09540261.2010.550868. PMID 21521086
- [Background] Lewis MA, Neighbors C, Oster-Aaland L, Kirkeby BS, Larimer ME. Indicated prevention for incoming freshmen: personalized normative feedback and high-risk drinking. Addict Behav. 2007 Nov;32(11):2495-508. doi: 10.1016/j.addbeh.2007.06.019. Epub 2007 Jun 28. PMID 17658695
- [Background] Neighbors C, Larimer ME, Lewis MA. Targeting misperceptions of descriptive drinking norms: efficacy of a computer-delivered personalized normative feedback intervention. J Consult Clin Psychol. 2004 Jun;72(3):434-47. doi: 10.1037/0022-006X.72.3.434. PMID 15279527
- [Background] Jacobson IG, Ryan MA, Hooper TI, Smith TC, Amoroso PJ, Boyko EJ, Gackstetter GD, Wells TS, Bell NS. Alcohol use and alcohol-related problems before and after military combat deployment. JAMA. 2008 Aug 13;300(6):663-75. doi: 10.1001/jama.300.6.663. PMID 18698065
- [Background] Sayer NA, Noorbaloochi S, Frazier P, Carlson K, Gravely A, Murdoch M. Reintegration problems and treatment interests among Iraq and Afghanistan combat veterans receiving VA medical care. Psychiatr Serv. 2010 Jun;61(6):589-97. doi: 10.1176/ps.2010.61.6.589. PMID 20513682
- [Background] Larimer ME, Turner AP, Mallett KA, Geisner IM. Predicting drinking behavior and alcohol-related problems among fraternity and sorority members: examining the role of descriptive and injunctive norms. Psychol Addict Behav. 2004 Sep;18(3):203-12. doi: 10.1037/0893-164X.18.3.203. PMID 15482075
- [Background] Lewis MA, Litt DM, Blayney JA, Lostutter TW, Granato H, Kilmer JR, Lee CM. They drink how much and where? Normative perceptions by drinking contexts and their association to college students' alcohol consumption. J Stud Alcohol Drugs. 2011 Sep;72(5):844-53. doi: 10.15288/jsad.2011.72.844. PMID 21906511
- [Background] Frone MR. Predictors of overall and on-the-job substance use among young workers. J Occup Health Psychol. 2003 Jan;8(1):39-54. doi: 10.1037//1076-8998.8.1.39. PMID 12553528
- [Background] McGonagle KA, Kessler RC. Chronic stress, acute stress, and depressive symptoms. Am J Community Psychol. 1990 Oct;18(5):681-706. doi: 10.1007/BF00931237. PMID 2075897
- [Background] Toker S, Biron M. Job burnout and depression: unraveling their temporal relationship and considering the role of physical activity. J Appl Psychol. 2012 May;97(3):699-710. doi: 10.1037/a0026914. Epub 2012 Jan 9. PMID 22229693
- [Background] Brown GP, Hammen CL, Craske MG, Wickens TD. Dimensions of dysfunctional attitudes as vulnerabilities to depressive symptoms. J Abnorm Psychol. 1995 Aug;104(3):431-5. doi: 10.1037//0021-843x.104.3.431. PMID 7673566
- [Background] Finlay-Jones R, Brown GW. types of stressful life event and the onset of anxiety and depressive disorders. Psychol Med. 1981 Nov;11(4):803-15. doi: 10.1017/s0033291700041301. PMID 7323236
- [Background] Lewis MA, Neighbors C. Optimizing personalized normative feedback: the use of gender-specific referents. J Stud Alcohol Drugs. 2007 Mar;68(2):228-37. doi: 10.15288/jsad.2007.68.228. PMID 17286341
- [Background] Geisner IM, Neighbors C, Larimer ME. A randomized clinical trial of a brief, mailed intervention for symptoms of depression. J Consult Clin Psychol. 2006 Apr;74(2):393-9. doi: 10.1037/0022-006X.74.2.393. PMID 16649884